CLINICAL TRIAL: NCT01477138
Title: Comparison of Right Ventricular Septal Pacing to Minimized Right Ventricular Septal Stimulation in Patients With Sick Sinus Syndrome
Brief Title: RV Septal Versus Minimized RV Pacing in Sick Sinus Syndrome
Acronym: VOTE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Klinikum Nürnberg (Other)
Responsible Party: Principal Investigator, Natalia Rohr, Natalia Rohr, Klinikum Nürnberg
Other Study IDs: VOTEPM
Record Dates: First submitted 2011-07-05; First posted 2011-11-22 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Sick Sinus Syndrome
Keywords: Sick Sinus Syndrome; Cardiac Pacing, Artificial; Cardiac Resynchronization Therapy; Pacemaker, Artificial; SSS
MeSH Terms: conditions — Sick Sinus Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- DDD(R): SSS. PM programmed to DDD(R) mode with ventricular pacing on the right ventricular septum.
  Interventions: Procedure: pacemaker implantation, AAI(R)-DDD(R) versus DDD(R)
- AAI(R)<=>DDD(R): SSS, PM-mode programmed for minimizing right ventricular pacing on the right interventricular septum
  Interventions: Procedure: pacemaker implantation, AAI(R)-DDD(R) versus DDD(R)

INTERVENTIONS:
Procedure: pacemaker implantation, AAI(R)-DDD(R) versus DDD(R) — Indication for pacemaker implantation: sick sinus syndrome in conformity with the current guidelines. Only market-released CE certified 2-chamber cardiac pacemakers and electrodes are used. The implantation is done according to the applicable standards. Active RV-lead is positioned on the right ventricular septum.
  Other Names: AAI(R)<=>DDD(R); DDD(R)

SUMMARY:
Background:

* Potential negative effects of pacing in the RV-apex are well documented
* However, study results comparing septal / RVOT-pacing versus RV-apical pacing controversial.
* The optimal pacing mode in SSS (DDDR versus AAIR) is unclear, as the DDD (R) mode with an AV delay ≤ 220 ms should be the preferred pacing mode, according to the DANPACE trial [DANPACE, ESC 2010, Stockholm].

Aim:

- to evaluate chronic effects of proven right ventricular septal compared to minimized right ventricular septal pacing in patients with SSS

Inclusion criterion:

-Pacemaker indication according to current guidelines: sick sinus syndrome (SSS)

Exclusion criteria:

* Life expectancy < 2 years
* Age <18 years
* Noncompliance with regard to participation in the study
* Pregnancy
* AV block ° 2 and higher
* Permanent atrial fibrillation
* Heart failure NYHA III and IV, reduced LV-EF <40%
* ICD indication
* Acute coronary syndrome. PCI or CABG <3 months
* Heart transplant
* Placement of septal RV electrode is not possible

Study design:

* Prospective, monocentric, randomized, double-blinded
* Run-in phase: for weeks AAI [R]-DDD [R]
* Randomization: two groups A) septal right ventricular chamber pacing: mode DDD [R] versus B) Reduction of unnecessary ventricular pacing: AAI [R]-DDD [R].
* FU: 6 and 12-months

Primary endpoints:

-LV ejection fraction and end-systolic LV volume after 12 months.

Secondary endpoints:

-LV end-diastolic volume, TAPSE, parameters of dyssynchrony (SPWMD, LV-PEP, IVMD), AF-burden, % ventricular pacing, CPX: peak oxygen consumption (peak VO2), VO2 AT, VO2/HR, VE/VCO2 slope; QoL scores (SF-36) after 12 months.

Statistics/sample size estimation:

In order to detect a difference in LVEF of 5% and for LV-ESV of 5 mL between the 2 groups after 12 months:

* 90% power/alpha 5%: 84 patients per group
* 80% power/alpha 5%: 63 patients per group

  * 10% for compensation of drop-outs / patients lost of follow-up. Two-sided 5% type 1 error Analysis intention-to-treat and based on the finally programmed pacing mode.

Material

* PG: market released dual chamber pacemakers with the ability to pace AAI(R) -DDD(R)
* pacing leads: market-released standard active electrodes
* RV electrode: septal verified under multi-level screening (RAO/LAO) and ECG (LBBB narrow <150 ms / inferior axis)

DETAILED DESCRIPTION:
Background:

* Potential negative effects of pacing in the RV-apex are well documented
* Asynchronous ventricular activation
* reduction of systolic and diastolic LV function
* Experimental data: histological changes
* Asymmetric LV hypertrophy and thinning
* However, study results comparing septal / RVOT-pacing versus RV-apical pacing controversial:
* Acute versus chronic
* Small number of cases, uncontrolled, unblinded,
* Brief periods of observation in the cross-over design (3 months)
* "RVOT" often summarizes different stimulation sites: high RVOT, lateral, septal. Actually only limited data with proven septal stimulation
* No objective performance assessment (CPX)
* Assessment of alternative stimulation site previously RVOT versus RV-apex,
* ventricular pacing compared to ventricular pacing, then tested a potential harm to another
* The question of the optimal pacing mode of patients with SSS (DDDR versus AAIR) appears to be open again. While in Germany, two-chamber systems with AAI [R] mode with ventricular back-up are used, should the DDD (R) mode with an AV delay ≤ 220 ms be the preferred pacing mode, according to the results of the DANPACE trial for patients with SSS [DANPACE, ESC 2010, Stockholm].

Aim:

- to evaluate chronic effects of proven right ventricular septal compared to minimized right ventricular septal pacing in patients with SSS

Inclusion criterion:

-Pacemaker indication according to current guidelines: sick sinus syndrome (SSS)

Exclusion criteria:

* Life expectancy < 2 years
* Age <18 years
* Noncompliance with regard to participation in the study
* Pregnancy
* AV block ° 2 and higher
* Permanent atrial fibrillation
* Heart failure NYHA III and IV, reduced LV-EF <40%
* ICD indication
* Acute coronary syndrome. PCI or CABG <3 months
* Heart transplant
* Placement of septal RV electrode is not possible

Study design:

* Prospective, monocentric, randomized, double-blinded
* Run-in phase: 4 weeks AAI [R]-DDD [R]
* ECG, PM-interrogation, echocardiography, performance diagnostics, CPX, QoL questionnaire
* Randomization: two groups 4 weeks (between 3 to 6 weeks) after implant A) septal right ventricular chamber pacing: mode DDD [R] versus B) Reduction of unnecessary ventricular pacing: AAI [R]-DDD [R].
* FU: 6 and 12-months
* ECG, Holter-ECG, PM-interrogation, echocardiography, performance diagnostics, CPX, QoL questionnaire
* Extension of follow-up if possible

Primary endpoints:

-LV ejection fraction and end-systolic LV volume after 12 months.

Secondary endpoints:

-LV end-diastolic volume, TAPSE, parameters of dyssynchrony (SPWMD, LV-PEP, IVMD), AF-burden, % ventricular pacing, CPX: peak oxygen consumption (peak VO2), VO2 AT, VO2/HR, VE/VCO2 slope; QoL scores (SF-36) after 12 months.

Blinding:

* Patient compared to the pacing mode
* Physician: offline analysis of echo and CPX blinded to the pacing mode

Statistics/sample size estimation:

In order to detect a difference in LVEF of 5% and for LV-ESV of 5 mL between the 2 groups after 12 months:

* 90% power/alpha 5%: 84 patients per group
* 80% power/alpha 5%: 63 patients per group

  * 10% for compensation of drop-outs / patients lost of follow-up. Two-sided 5% type 1 error Analysis intention-to-treat and based on the finally programmed pacing mode.

Material

* PG: market released dual chamber pacemakers with the ability to pace AAI(R) -DDD(R)
* pacing leads: market-released standard active electrodes (eg. BSCI FineLine 4470 and 4471) Implantation
* Transvenously
* RA-electrode: if possible, short atrial conduction time
* RV electrode: septal verified under multi-level screening (RAO/LAO) and ECG (LBBB narrow <150 ms / inferior axis)

ELIGIBILITY:
Inclusion Criteria:

* Pacemaker indication according to current guidelines: sick sinus syndrome (SSS)

Exclusion Criteria:

* Life expectancy <2 years
* Age < 18 years
* Noncompliance with regard to participation in the study
* Pregnancy
* AV block ° 2 and higher
* Permanent atrial fibrillation
* Heart failure NYHA III and IV, reduced LV-EF < 40%
* ICD indication
* Acute coronary syndrome. PCI or CABG < 3 months
* Heart transplant
* Placement of septal RV electrode is not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with symptomathic sick sinus syndrome
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
end-systolic LV volume | at randomisation and after 12 months
left ventricular ejection fraction (LV-EF) | at randomisation and after 12 months
  TTE, Simpson, biplane

SECONDARY OUTCOMES:
TAPSE | at randomisation and after 12 months
echocardiographic parameter of dyssynchrony | at randomisation and after 12 months
  TTE, SPWMD, LV-PEP, IVMD
peak VO2, VO2 AT, VO2/HR, VE/VCO2 slope | at randomisation and after 12 months
  CPX: cardiopulmonary exercice testing
quality of life-scores | at randomisation and after 12 months
  SF-36
AF burden | at randomisation and after 12 months
% ventricular pacing | at randomisation and after 12 months
LV end diastolic volume | at randomisation and after 12 months
  TTE

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Pauschinger, Prof.Dr.med., Study Chair — Klinikum Nuernberg South/ Cardiology; Dirk Bastian, MD, Principal Investigator — Klinikum Nuernberg
Locations (1):
- Klinikum Nuernberg South, Nuremberg, Bavaria, Germany

REFERENCES:
- [Background] Schwaab B, Frohlig G, Alexander C, Kindermann M, Hellwig N, Schwerdt H, Kirsch CM, Schieffer H. Influence of right ventricular stimulation site on left ventricular function in atrial synchronous ventricular pacing. J Am Coll Cardiol. 1999 Feb;33(2):317-23. doi: 10.1016/s0735-1097(98)00562-2. PMID 9973009
- [Background] Tse HF, Yu C, Wong KK, Tsang V, Leung YL, Ho WY, Lau CP. Functional abnormalities in patients with permanent right ventricular pacing: the effect of sites of electrical stimulation. J Am Coll Cardiol. 2002 Oct 16;40(8):1451-8. doi: 10.1016/s0735-1097(02)02169-1. PMID 12392836
- [Background] Sweeney MO, Hellkamp AS, Ellenbogen KA, Greenspon AJ, Freedman RA, Lee KL, Lamas GA; MOde Selection Trial Investigators. Adverse effect of ventricular pacing on heart failure and atrial fibrillation among patients with normal baseline QRS duration in a clinical trial of pacemaker therapy for sinus node dysfunction. Circulation. 2003 Jun 17;107(23):2932-7. doi: 10.1161/01.CIR.0000072769.17295.B1. Epub 2003 Jun 2. PMID 12782566
- [Background] Wilkoff BL, Cook JR, Epstein AE, Greene HL, Hallstrom AP, Hsia H, Kutalek SP, Sharma A; Dual Chamber and VVI Implantable Defibrillator Trial Investigators. Dual-chamber pacing or ventricular backup pacing in patients with an implantable defibrillator: the Dual Chamber and VVI Implantable Defibrillator (DAVID) Trial. JAMA. 2002 Dec 25;288(24):3115-23. doi: 10.1001/jama.288.24.3115. PMID 12495391
- [Background] Stambler BS, Ellenbogen K, Zhang X, Porter TR, Xie F, Malik R, Small R, Burke M, Kaplan A, Nair L, Belz M, Fuenzalida C, Gold M, Love C, Sharma A, Silverman R, Sogade F, Van Natta B, Wilkoff BL; ROVA Investigators. Right ventricular outflow versus apical pacing in pacemaker patients with congestive heart failure and atrial fibrillation. J Cardiovasc Electrophysiol. 2003 Nov;14(11):1180-6. doi: 10.1046/j.1540-8167.2003.03216.x. PMID 14678131
- [Background] Giudici MC, Thornburg GA, Buck DL, Coyne EP, Walton MC, Paul DL, Sutton J. Comparison of right ventricular outflow tract and apical lead permanent pacing on cardiac output. Am J Cardiol. 1997 Jan 15;79(2):209-12. doi: 10.1016/s0002-9149(96)00718-7. PMID 9193029
- [Background] de Cock CC, Meyer A, Kamp O, Visser CA. Hemodynamic benefits of right ventricular outflow tract pacing: comparison with right ventricular apex pacing. Pacing Clin Electrophysiol. 1998 Mar;21(3):536-41. doi: 10.1111/j.1540-8159.1998.tb00095.x. PMID 9558684
- [Background] Alboni P, Scarfo S, Fuca G, Mele D, Dinelli M, Paparella N. Short-term hemodynamic effects of DDD pacing from ventricular apex, right ventricular outflow tract and proximal septum. G Ital Cardiol. 1998 Mar;28(3):237-41. PMID 9561877
- [Background] Yu CM, Chan JY, Zhang Q, Omar R, Yip GW, Hussin A, Fang F, Lam KH, Chan HC, Fung JW. Biventricular pacing in patients with bradycardia and normal ejection fraction. N Engl J Med. 2009 Nov 26;361(22):2123-34. doi: 10.1056/NEJMoa0907555. Epub 2009 Nov 15. PMID 19915220
- [Result] Nielsen, Jens Cosedis - Blomstrom-Lundqvist, Carina. DANPACE: The Danish multicenter randomised trial on single lead atrial versus dual chamber pacing in sick sinus syndrome. ESC Kongress 2010, Stockholm, Session number: 708001 - 70800.